CLINICAL TRIAL: NCT05853042
Title: MERITnI - Mindray-hs-cTnI Assay: Analytical and Clinical Evaluation for the Diagnosis and RIsk AssessmenT of Myocardial InfarctIon.
Acronym: MERITnI
Status: Active, not recruiting | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Mindray Bio-Medical Electronics Co., Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: MERITnI
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction; Acute Coronary Syndrome
Keywords: cardiac troponin; acute myocardial injury; acute myocardial infarction; high-sensitivity cardiac troponin I; Mindray; Mindray Bio-medical; Cardiac troponin I; Reference range; Abbott Alinity; Type 1 myocardial infarction; Type 2 myocardial infarction; Risk outcomes assessment
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiomyopathy, Dilated, 1FF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples tested on the Mindray Bio-Medical CL-1200i Chemiluminescence Immunoassay Analyzer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Study population: Prospective, observational cohort study of consecutive patients (goal, 1500 patients over 4 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
  Interventions: Diagnostic Test: high-sensitivity cardiac troponin testing

INTERVENTIONS:
Diagnostic Test: high-sensitivity cardiac troponin testing — Lithium heparin plasma samples will be measured with Mindray Bio-Medical CL-1200i Chemiluminescence Immunoassay Analyzer.

SUMMARY:
The Mindray High Sensitivity Troponin-I Measurement System is an in vitro diagnostic test for the quantitative determination of high sensitivity cardiac troponin I (hs-cTnI) in human serum or plasma.

The Mindray High Sensitivity Troponin-I Measurement System is to be used as an aid in the diagnosis and rule out of acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
Study purpose/objective:

* Determine the sex-specific 99th percentile upper reference limits (URLs) for the Mindray hs-cTnI assay using the CL-1200i Instrument.
* Method comparison across the dynamic range of cTnI concentrations between the Mindray hs-cTnI assay and the Abbott Alinity hs-TnI assay used in clinical practice at Hennepin Healthcare/Hennepin County Medical Center.
* Evaluate the clinical performance of the Mindray hs- cTnI measuring system for the diagnosis of myocardial infarction (MI), for early rule out MI and myocardial injury, and assessment of 30-day safety outcomes in patients presenting to the emergency department (ED) in whom serial cTnI measurements (0h, 2h, 4h, 6h) are obtained on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN USA) to rule-in and rule-out MI.

ELIGIBILITY:
Inclusion Criteria:

1. Presents to the ED, or ambulatory care center equivalent, with signs or symptoms suspicious of a possible ACS/ischemic event.
2. Baseline cTn-I measurement and one additional cTn-I measurement at two hours after the first measurement.
3. At least one 12-lead electrocardiogram

Exclusion Criteria:

1. Less than 21 years old
2. Pregnancy
3. Trauma
4. Declines to participate or has indicated that their blood/ medical information cannot be used for investigational purposes
5. Did not present through the ED
6. Transferred from an outside hospital or clinic
7. Has already been enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients (goal, 1500 patients over 4 months) presenting to the emergency department, in whom serial cTnI measurements are ordered on clinical indication at Hennepin Healthcare / Hennepin County Medical Center (Minneapolis, MN, USA) to rule-in and rule-out acute myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Examine the incidence of undetectable(<LoD), measurable (LoD - 99th percentile), and increased (>99th percentile) cTn concentrations for the Mindray Bio-Medical hs-cTnI assay using the CL-1200i analyzer. | Day 1
  Examine the incidence of undetectable(<LoD), measurable (LoD - 99th percentile), and increased (>99th percentile) cTn concentrations for the Mindray Bio-Medical hs-cTnI assay using the CL-1200i analyzer in comparison to a high sensitivity cTnI assay (Abbott Alinity) to determine the potential impact on positivity rate, defined by sex-specific 99th percentiles.
Examine Concordance | Day 1
  Examine analytical and clinical concordance and discordance predicated on sex-specific 99th percentiles between Mindray hs-cTnI concentrations in comparison to the Abbott Alinity high sensitivity cTnI assay.
Examine the diagnostic performance for acute myocardial injury and acute myocardial infarction. | Day 1
  Examine the diagnostic performance for a) acute myocardial injury and b) acute myocardial infarction based on various diagnostic strategies using hs-cTnI measurement(s), as follows:
  1. Single measurement rule out strategy
     1. Limit of detection (LoD)
     2. Derive an optimal rule-out (ng/L) hs-cTnI cutoff for the Mindray Bio-Medical hs-cTnI assay using the CL-1200i analyzer to meet an early rule out clinical need
  2. Accelerated serial sampling (0/2h protocol) rule out strategy
     a) Delta (absolute concentration serial change value, 0-2h) analysis
  3. Diagnosis performance predicated on sex-specific 99th percentile URLs
Describe the incidence of MI and myocardial injury, clinical characteristics and 30-day safety outcomes risk of patients with and without hs-cTnI increases above the sex-specific 99th percentile URLs | Day 1
  Describe the incidence of MI and myocardial injury, clinical characteristics and 30-day safety outcomes risk of patients with and without hs-cTnI increases above the sex-specific 99th percentile URLs, including patients categorized with acute myocardial injury and acute myocardial infarction, including type 1 and 2 myocardial infarction, following the 4th Universal Definition of Myocardial Infarction.
Impact on the incidence of myocardial injury and myocardial infarction diagnoses. | Day 1
  Examine the potential impact on the incidence of myocardial injury and myocardial infarction diagnoses using hs-cTnI upon clinical practice implementation with a comparison to the hospital's final ICD-10 code diagnosis of type 1 and type 2 MIs, and non-MI myocardial injury.

SECONDARY OUTCOMES:
All-cause mortality | up to 30 days
  All cause death
Cardiac mortality | up to 30 days
  Death due to cardiac pathophysiology
Adjudicated index acute myocardial infarction according to Fourth Universal Definition of Myocardial Infarction. | on admission
  Acute myocardial infarction including all sub-types following the Fourth Universal Definition of Myocardial Infarction guidelines.
Safety Outcomes | 30 days
  Determine major adverse cardiovascular events, including cardiac death, myocardial infarction, unplanned revascularization and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Fred S Apple, PhD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare Research Institute / Hennepin County Medical Center, Minneapolis, Minnesota, United States